CLINICAL TRIAL: NCT06898710
Title: Evaluating the Efficacy of Patient Specific Z-shape Mini-plate With Lingual Extension Versus Usual Two Mini-plates in Mandibular Class III Fracture Management
Brief Title: z Mini-plate With Lingual Extension Versus Conventional 2 Mini Plates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, associate professor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4444
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Mandible Fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- z miniplate with lingual extension (Experimental)
  Interventions: Procedure: z mini plate with lingual extension
- two mini plate (Active Comparator)
  Interventions: Procedure: conventional 2 mini plates

INTERVENTIONS:
Procedure: z mini plate with lingual extension — patient with class III mandible fracture will be treated with patient specific z mini plate with lingual extension
  Arms: z miniplate with lingual extension
Procedure: conventional 2 mini plates — patient with class III mandible fracture will be treated with conventional 2 mini plates
  Arms: two mini plate

SUMMARY:
The collected patients according to the eligibility criteria will be randomly distributed into one of these groups:

Group I : 10 patients suffering class III mandibular fracture will be managed by patient specific Z shape mini-plate with lingual extension (study group).

Group II : 10 patients suffering class III mandibular fracture will be managed by 2 mini plates at superior and inferior borders (control group).

The allocation sequence will be generated using computerized random numbers and kept in sealed envelopes, which will be opened prior to surgery. All patients will provide the informed consent after declaration the procedures, benefits, and harms

ELIGIBILITY:
Inclusion Criteria:

* - Class III mandibular fracture
* medically stable patient
* aged above 21 years
* no medical condition affect the bone healing

Exclusion Criteria:

* • absence of other facial trauma, mandibular condylar fracture

  * patient refuse the follow up

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
inter condylar distance | 3 months

IPD SHARING:
Plan to Share IPD: Undecided